CLINICAL TRIAL: NCT04046718
Title: Lipid Profile Response to Electroacupuncture
Brief Title: Lipid Profile Response to Electroacupuncture Stimulation in Non Alcoholic Fatty Liver Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramy Salama Draz (Other)
Responsible Party: Sponsor-Investigator, Ramy Salama Draz, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/001579_1
Record Dates: First submitted 2019-08-03; First posted 2019-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Fatty Liver , Electroacupuncture, Lipid Profile
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Intervention Model Description: two group study, one is the study group and the other is a control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupuncture (Experimental): the study group received electroacupuncture stimulation at different points
  Interventions: Device: electro-acupuncture stimulation
- control group (No Intervention): a control group with no intervention

INTERVENTIONS:
Device: electro-acupuncture stimulation — stimulation of acupoints of the liver meridian of lv3 lv14
  Arms: electroacupuncture

SUMMARY:
sixty female patients suffering from non-alcoholic fatty liver disease were randomly divided into two equal groups group 1 received electroacupuncture stimulation for 6 weeks at special points of stimulation. group 2 was a control group that received nothing without any change in lifestyle and we assed the response of lipid profile post-treatment protocol in both groupes

ELIGIBILITY:
Inclusion Criteria:

non alcoholic fatty liver BMI 30-40

Exclusion Criteria:

* Patients with: (Hepatitis C & b any form of seizure

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-12-29 (Actual)

PRIMARY OUTCOMES:
tri-triglycerides (mg/dl) , total cholesterol (mg/dl) , HDL (mg/dl) , LDL (mg/dl) | 6 weeks
  lowering of total lipid profile in study group

SECONDARY OUTCOMES:
weight (kg) , height (m), BMI (kg/m2) | 1st week
  calculation of body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Draz RS, Serry ZMH, Rahmy AF, El Bardesi MS, Taha MM. Electroacupuncture Versus Aerobic Interval Training on Liver Functions in Patients with Nonalcoholic Fatty Liver. J Altern Complement Med. 2020 Jan;26(1):51-57. doi: 10.1089/acm.2019.0182. Epub 2019 Oct 29. PMID 31657614
- See also: my orcid account ID — https://orcid.org/0000-0003-4089-323X